CLINICAL TRIAL: NCT00883805
Title: Investigation of Systemic Metal Ion Concentration Following a Ceramic-on-metal Total Hip Arthroplasty
Status: Withdrawn | Type: Observational
Why Stopped: PI moved
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Daniel Grande, director:orthopaedic research, Northwell Health
Other Study IDs: GCRC 0163; IRB# 07-08-105
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Hip Replacement; Hip Implant; Total Hip Arthroplasty; Orthopaedic Surgery
Keywords: Metal Ion Concentration; Osteolysis
MeSH Terms: conditions — Osteolysis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Metal-on-Metal Articulations: Subjects will be people who have had metal-on-metal total hip arthroplasties
  Interventions: Biological: Blood draw; Radiation: X-Ray of Hip
- Ceramic-on-Metal Articulations: Subjects will be people who have had ceramic-on-metal total hip arthroplasties
  Interventions: Biological: Blood draw; Radiation: X-Ray of Hip

INTERVENTIONS:
Biological: Blood draw — Subjects will give blood for analysis of metal ion concentrations
Radiation: X-Ray of Hip — Subject will have x-ray of hip to assessment of osteolysis

SUMMARY:
This is a pilot study to compare systemic concentrations of cobalt and chromium in patients that have previously undergone total hip arthroplasties with ceramic on metal and metal on metal bearing surfaces.

DETAILED DESCRIPTION:
This is a pilot study to compare systemic concentrations of cobalt and chromium in patients that have previously undergone total hip arthroplasties with ceramic on metal and metal on metal bearing surfaces. Secondary goals include an assessment of osteolysis on radiographs, potential long term analysis of implant survivability, and cancer rates in the two patient populations.

Increased metal ion production has been documented in metal-on-metal arthroplasty articulations. There are several concerns over metal ion production. First, even though there is a decreased histiocytic response to metallic debris, a dose dependent cytotoxic response with Interleukin 6, Prostaglandin E2, and Tumor Necrosis Factor alpha persists and may cause osteolysis in the long term. Second, increased levels of cobalt, chromium and nickel has been shown to correlate with increased cancer rates in several animal models, and the carcinogenic risk in humans has not been fully elucidated as yet. Third, hypersensitivity reactions to metal ion develop in up to 25% of these patients, and 60% of patients with poorly functioning hip.

Ceramic on metal avoids many of these problems due to the improved wear characteristics. If the level of metal ion production is significantly reduced and the implant survivability is proven in long term studies, this articulation may become the preferred method.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 40 - 80, who has undergone a top hip arthroplasty with either metal on metal or ceramic on metal articulation for a diagnosis of non-inflammatory degenerative joint disease. We will also include subjects who have had bilateral hip arthroplasties or a second arthroplasty performed since the initial surgery.
* Patient must be able to provide consent to participate

Exclusion Criteria:

* Diagnosis other than non-inflammatory degenerative joint disease, chronic renal insufficiency, or any systemic inflammatory condition
* Evidence of active infections
* Patients whose occupations include welding or metal working
* A second arthroplasty performed since the initial will not be exclude, but their data will be analyzed as a subpopulation
* unwillingness to comply with rehabilitation program or inability to return for follow-up visits
* Any systemic steroid therapy within 3 months of surgery
* Subjects who are pregnant

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled will have already undergone a total hip arthroplasty with either a metal-on-metal articulation, or a ceramic-on-metal articulation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
metal ion concentration in urine | 1 year post-op

SECONDARY OUTCOMES:
metal ion concentration in blood | 1 year post-op

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Grande, Ph.D., Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States